CLINICAL TRIAL: NCT03806205
Title: Efficacy Management and Adherence Evaluation of Diclofenac in the Treatment of Knee Osteoarthritis Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PekingUPHmed
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: To Investigate the Effect of Diclofenac on Pain Control of Knee Osteoarthritis and the Relationship Between Pain Relief and Medicine Adherence
Keywords: Knee osteoarthritis pain; Adherence; Diclofenac; Follow up
MeSH Terms: interventions — Organization and Administration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: regular follow-up — we give a regular follow-up and supervision on the study group
  Other Names: supervision

SUMMARY:
To investigate the effect of dichloride on pain control of knee osteoarthritis and the relationship between pain relief and medicine adherence. To evaluate the pain relief rate of patients with different initial pain.

ELIGIBILITY:
Inclusion Criteria:

* According to the OA diagnostic criteria of knee joint, the side with higher WOMAC score is defined as observing knee joint for patients with both knees conforming to OA diagnostic criteria.

  1. Repeated knee pain in the past month
  2. X-ray showed narrowing of articular space, subchondral sclerosis and/or cystic degeneration, and formation of osteophyte at articular margin.
  3. Joint fluid (> 2 times) is cool and sticky, WBC < 2000/ml
  4. Age over 40
  5. Morning stiffness less than 30 minutes
  6. Bone fricative (sensation) during exercise According to 1+2 or 1+3+5+6 or 1+4+5+6, OA of knee joint can be diagnosed.
  7. The informed consent has been signed

Exclusion Criteria:

* (1) Joint pain caused by other causes (infection, hip, lumbar and other diseases) (2) Secondary arthritis (rheumatoid arthritis, ankylosing spondylitis, etc.) (3) Severe internal medical complications and other inability to participate in the research (4) Pain in other parts exceeds joint pain (5) Contraindications to diclofenac use: active peptic ulcer/allergy/induced asthma (6) Assessment may not complete the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-15 (Estimated); Primary Completion 2019-03-10 (Estimated); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
adherence | 6-8 weeks
  We will calculate adherence with medication use
pain relief rate | 6-8 weeks
  We will calculate the pain relief rate on all participants

SECONDARY OUTCOMES:
womac score | 6-8 weeks
  We will calculate the womac score on all participants

CONTACTS AND LOCATIONS:
Overall Officials: Jianhao Lin, M.D., Study Chair — Peking University People's Hospital; Yudian Qiu, M.D., Study Director — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Xicheng District, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] da Costa BR, Reichenbach S, Keller N, Nartey L, Wandel S, Juni P, Trelle S. RETRACTED: Effectiveness of non-steroidal anti-inflammatory drugs for the treatment of pain in knee and hip osteoarthritis: a network meta-analysis. Lancet. 2016 May 21;387(10033):2093-2105. doi: 10.1016/S0140-6736(16)30002-2. Epub 2016 Mar 18. PMID 26997557 (Retraction: PMID 28699579 Lancet. 2017 Jul 8;390(10090):109)